CLINICAL TRIAL: NCT03238716
Title: Neuromuscular Re-education, Impairment-based Exercise and Electric Dry Needling vs. Neuromuscular Re-education and Impairment-based Exercise for Stress Urinary Incontinence
Brief Title: Neuromuscular Re-eduaction, Exercise and Electric Dry Needling vs. Neuromuscular Re-education and Exercise for Stress Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit an adequate number of patients with stress urinary incontinence (based on inclusion / exclusion criteria) to participate in the study
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Primary Investigator and President of Spinal Manipulation Institute and Dry Needling Institute of the American Academy of Manipulative Therapy, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0015
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric DN, NM Re-ed, Exercise (Experimental)
  Interventions: Other: Electric DN; Other: NM Re-ed; Other: Exercise
- NM Re-ed and Exercise (Active Comparator)
  Interventions: Other: NM Re-ed; Other: Exercise

INTERVENTIONS:
Other: Electric DN — Dry needling with electric stimulation to the erector spine and paraspinal muscles in the lumbar / sacral region and tibialis anterior / posterior. Dry needling with electric stimulation of peri-neural tissue associated with lumbar / sacral nerve roots, pudendal nerve and posterior tibial nerve. 8-12 treatment sessions over 6 weeks.
  Arms: Electric DN, NM Re-ed, Exercise
Other: NM Re-ed — sEMG targeting type I slow-twitch fibers and type II fast-twitch fibers. Type I fibers maintain continuous muscle activity over prolonged periods of time; therefore, training of type I fibers will be achieved through endurance and repetition training of the pelvic floor muscles. Type II fibers are recruited during sudden increases in intra-abdominal pressure, and these fibers will be recruited with "The Knack" training. The Knack is a term created to use rhythm or timing to the pelvic floor. Neuromuscular re-education will be performed during the first treatment, but it will be performed "as needed" on subsequent treatments.
Other: Exercise — Impairment-specific strength training, which may include transversus abdominis (TrA), gluteus maximus/medius/minimus and/or hip abductor/adductor muscle training. Treadmill, riding the recumbent bike at > 2 METs and/or stair climbing. Exercise training will be performed 7-11 treatment sessions over 6 weeks (following treatment 1).

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with stress urinary incontinence: neuromuscular re-education, impairment-based exercise and electric dry needling versus neuromuscular re-education and impairment-based exercise. Physical therapists commonly use all of these techniques to treat stress urinary incontinence. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with stress urinary incontinence will be randomized to receive 2 treatment sessions per week for up to 6 weeks (8-12 sessions total) of either: (1) neuromuscular re-education, impairment-based exercise and electric dry needling (2) neuromuscular re-education and impairment-based exercise

ELIGIBILITY:
Inclusion Criteria:

1. Aged 35 - 75 years
2. Female
3. Meet the diagnosis of stress urinary incontinence - urine leakage with increased abdominal pressure from laughing, sneezing, coughing, or other physical stressors on abdominal cavity and bladder

Exclusion Criteria:

1. Urge urinary incontinence or mixed urinary incontinence
2. Greater than second degree prolapse
3. Previous surgical intervention related to female anatomy
4. Urinary tract infection
5. Unable to participate in movement such as walking, stair climbing, or resistance training
6. Taking medication that impacts bladder function
7. Serious cardiovascular, cerebral disease, psychiatric disorder, cognitively impaired, injury of cauda equine, and/or myelopathy
8. Pregnancy
9. Sacral nerve stimulator implanted
10. Cardiac pacemaker, metal allergy, or severe needle phobia

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Incontinence Impact Questionnaire - Short Form IIQ-7 | baseline, 6 weeks, 3 months
  7 questions, each worth 0-3 points. The average score of items responded to is calculated, then multiplied by 33 1/3 to put the scores on a scale of 0 to 100. High scores indicate greater impact of incontinence.

SECONDARY OUTCOMES:
Global Rating of Change Scale | 6 weeks, 3 months
  15 point self-report scale (-7 to 7). High rating indicates a greater impact of change
Urinary pad per day usage | baseline, 6 weeks, 3 months
  Number of urinary pads that the patient requires per day secondary to stress urinary incontinence
Urogenital Distress Inventory | baseline, 6 weeks, 3 months
  6 questions, each worth 0-3 points. The raw score is divided by 6 then multiplied by 25 for the total score. High scores indicate more distress due to bladder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Research Physical Therapy Specialists, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided